CLINICAL TRIAL: NCT04334369
Title: Does Specialty Soft Contact Lens Wear Decrease the Onset and Progression of Myopia in Optometry School Interns?
Brief Title: Contact Lens and Myopia Control in Optometry School Students
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: LOSS OF FORMER PRINCIPAL INVESTIGATOR
Sponsor: Jeff Rabin (Other)
Responsible Party: Sponsor-Investigator, Jeff Rabin, PROFESSOR AND ASSISTANT DEAN, University of the Incarnate Word
Organization: University of the Incarnate Word (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RSO myopia control
Record Dates: First submitted 2020-03-26; First posted 2020-04-06 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2020-04

CONDITIONS: Myopia, Progressive
Keywords: Multifocal contact lenses; Myopia progression; Axial length
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Single Vision Contact Lenses (Sham Comparator)
  Interventions: Device: Proclear Single Vision Contact Lenses manufactured by CooperVision
- Multifocal Contact Lenses (Experimental)
  Interventions: Device: Proclear Multifocal Contact Lenses manufactured by CooperVision

INTERVENTIONS:
Device: Proclear Single Vision Contact Lenses manufactured by CooperVision — FDA approved single vision contact lenses.
  Arms: Single Vision Contact Lenses
Device: Proclear Multifocal Contact Lenses manufactured by CooperVision — FDA Approved Multifocal Contact Lenses
  Arms: Multifocal Contact Lenses

SUMMARY:
The purpose of the study is to determine the effect of Natural View Multifocal lenses, a soft multifocal lens, on retardation of myopia in an optometric student population. Close up work (i.e. reading, computer work, etc.) is thought to play a factor in the progression of myopia in young adults. The progression should be slowed if not stopped through the use of peripheral defocus lenses (Natural View Multifocal) to change the optics of the eye in order to focus the image on the peripheral retina as opposed to behind it.

DETAILED DESCRIPTION:
BACKGROUND AND SIGNIFICANCE Myopia is a common refractive error that has increased among young adults and has become more prevalent in the growing population across the globe (Fan, et al 2004). This has been more common in Eastern Asian countries with prevalence of myopia as high as 96.5% among 19 year old soldiers in South Korea. (Shimuzu, et al 2003) In the United States between the 1990's to the 2000's there was a sudden increase of >15% myopia progression (Vitale et al 2009). There has been a correlation between education and myopia progression in urban areas calling into question the amount of close up work and being indoors as opposed to being outside working as in the rural populations (Resnikoff, et al 2004). Children between the ages of 7 to 11 years that were forced to spend 80 minutes per day outside showed a significantly better outcome in regards to onset as well as progression of myopia. Those that were spending 80 minutes per day outside had an average onset of 8.4% and progression of 0.25 diopters whereas the children that were not forced to spend time outside had onset and progression at a rate of 17.7% and 0.38 diopters respectively. (Wu, et al 2013) Myopia progression has become a cause for concern due to the complications that arise from the elongation of the eye. Some of the complications include retinal detachment, choroidal thinning, glaucoma and myopic macular degeneration. In a study of the causes of visual impairment in an adult Chinese population, it was found that myopic macular degeneration was the leading cause of bilateral visual impairment in adults between the ages of 45 and 59 years old and the second highest major cause of bilateral blindness. (Tang Y, et al 2015) Pathological myopia is one of the leading causes of blindness that can be prevented (Kang et. al. 2017).

Recent studies have promising conclusions that soft multifocal contact lenses are a viable option for slowing myopia progression. Many studies have been conducted on the topic of myopic control with soft multifocal contact lenses in young patients. Very little data exists on myopia control methods used in young adults. It is often thought that myopic progression will progress even through to young adults which could potentially necessitate a need for control. If the use of Dual-Focus soft contact lenses in young adults controls myopia, this could become a viable, cost effective method to increase productivity around the world. This is an important factor to consider as the direct and indirect cost of loss of productivity due to uncorrected refractive error is 202 billion dollars. (WHO bulletin 2004). Reducing the negative side effects of myopia and possible reduced vision loss in this specific population can open doors to future research in other populations.

A common treatment for myopia progression is Orthokeratology, in which patients wear a rigid gas permeable contact lens overnight in the hope of reshaping their corneas. A major concern however, with this treatment is the increased risk of infection that comes with wearing a lens overnight. It is also not approved for use on patients with a refractive error of >6.00D of myopia, and is not effective in older adult patients (Cooper et al 2017). Another pitfall of Orthokeratology is that once treatment is stopped, the refractive error of the patient returns to normal. This treatment regimen is easily restricted due to the high cost to the patient. This in turn calls for a type of treatment that can be used during the day, is cost effective, and can be easily disposed of to decrease the risk of infection. If the daily multifocal soft contact lenses are used correctly, any risk of infection or major drawback is greatly reduced. Another method of treatment involves the use of Atropine, which has proven to be successful in controlling the advancement of myopia. This however has side effects including blurry vision, increased sensitivity to light, possible flushing, tachycardia, bradycardia and other undesirable side effects. As the dose of Atropine rises, the reported side effects also increase. (Huy et. al. 2017).

LOCATION, FACULTY AND EQUIPMENT TO BE USED

* University of Incarnate Word Rosenberg School of Optometry Eye and Vision Care Clinic
* IOL Master 500 by Zeiss
* Topography
* Pentacam

SUBJECTS AND INFORMED CONSENT

Ideal subjects should:

* Be first or second year Optometric students at RSO
* Be non-presbyopic
* Have at least -0.50 Diopters or more of myopia in one or both eyes
* Have no systemic health issues
* Have no previous history of Orthokeratology
* Have no gas permeable contact use in the last 6 months
* Not be enrolled in any other eye study
* Be able to have a cycloplegic refraction
* New and existing contact lens wearers An announcement will be made to the incoming and 2nd year classes in the classroom at the end of one of their lectures. Also a class wide email will be sent out to the 1st and 2nd years giving them the necessary information. A copy of the informers consent will be given for signature. Proper insertion and removal training will be given to new wearers.

DURATION Recruitment will cease within the first 2 months of the study. Data collection and analysis will be ongoing throughout the course of the study. The participants of this study will be monitored at 6 month intervals until their 4t h year of Optometry school.

TESTING Active time during each visit is about 30 minutes, potentially up to 60 minutes including inactive time. Through the use of the G-Power analysis we have decided that ideally 40 patients will be needed. All tasks will be provided by any available investigators or research staff, under necessary supervision.

One year visit : is a comprehensive exam (uncorrected VA, retinoscopy, refraction, cover test at distance and near with prism neutralization, extraocular motility, near point of convergence , amplitude of accommodation, pupil testing in bright and dim lighting, confrontation field, slit lamp exam with dry eye testing - sodium fluorescein staining and tear break up time) pentacam, A scan, cycloplegic refraction (cyclopentolate 1%), dilated fundus exam yearly, OCT.

Uncorrected VA, dry refraction, cyclo refraction, cover tests (Distance and near), amps, slit lamp exam with dry eye eval (TBUT, and sodium fluorescein test) , dilated eye exam, baseline macular OCT

Six month Visit: Comprehensive exam, consider cycloplegic refractions if at least a -0.50D myopic shift or more is suspected. A-Scan, topography, pentacam, visual comfort questionnaire also performed.

Risk Analysis: Bacterial keratitis, corneal neovascularization, dry eyes secondary to contact lens wear, ocular discomfort, potential allergic reactions contact lens solution. All subjects will be given a contact number should they experience any complications during the study.

ELIGIBILITY:
Inclusion Criteria:

* Be first or second year Optometric students at RSO
* Be non-presbyopic
* Have at least -0.50 Diopters or more of myopia in one or both eyes
* Have no systemic health issues
* Have no previous history of Orthokeratology
* Have no gas permeable contact use in the last 6 months
* Not be enrolled in any other eye study
* Be able to have a cycloplegic refraction
* New and existing contact lens wearers

Exclusion Criteria:

* Progressive retinal or corneal disorder as well as any of the above

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2022-07-03 (Actual); Study Completion 2022-07-03 (Actual)

PRIMARY OUTCOMES:
Contact Lenses and Myopia Progression | 3 years
  Changes in axial length in millimeters
Contact Lenses and Myopia Progression | 3years
  Progression of Myopia in Diopters

CONTACTS AND LOCATIONS:
Overall Officials: Mervyn Bloom, OD, Principal Investigator — University of the Incarnate Word
Locations (1):
- Bowden Eye Care & Health Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] D. Lee, Y. Pang, R. Patel, M. Patel. A study of myopia progression in young adults Investigate Ophthalmology and Vision Science: An ARVO Journal. 2008;49(13)
- [Background] Fedtke C, Ehrmann K, Holden BA. A review of peripheral refraction techniques. Optom Vis Sci. 2009 May;86(5):429-46. doi: 10.1097/OPX.0b013e31819fa727. PMID 19342977
- [Background] Kang P, McAlinden C, Wildsoet CF. Effects of multifocal soft contact lenses used to slow myopia progression on quality of vision in young adults. Acta Ophthalmol. 2017 Feb;95(1):e43-e53. doi: 10.1111/aos.13173. Epub 2016 Aug 6. PMID 27495880
- [Background] Multifocal contact lens effective at treating myopia in kids. American Optometric Association. April 25, 2016. Available from: https://www.aoa.org/news/clinical-eye-care/multifocal-contact-lens-effective-at-treating-myopia-in-kids.
- [Background] Walline JJ, Greiner KL, McVey ME, Jones-Jordan LA. Multifocal contact lens myopia control. Optom Vis Sci. 2013 Nov;90(11):1207-14. doi: 10.1097/OPX.0000000000000036. PMID 24061152
- [Background] Li SM, Ji YZ, Wu SS, Zhan SY, Wang B, Liu LR, Li SY, Wang NL, Wang JJ. Multifocal versus single vision lenses intervention to slow progression of myopia in school-age children: a meta-analysis. Surv Ophthalmol. 2011 Sep-Oct;56(5):451-60. doi: 10.1016/j.survophthal.2011.06.002. Epub 2011 Aug 2. PMID 21813146
- [Background] Fan DS, Lam DS, Lam RF, Lau JT, Chong KS, Cheung EY, Lai RY, Chew SJ. Prevalence, incidence, and progression of myopia of school children in Hong Kong. Invest Ophthalmol Vis Sci. 2004 Apr;45(4):1071-5. doi: 10.1167/iovs.03-1151. PMID 15037570
- [Background] Shimizu N, Nomura H, Ando F, Niino N, Miyake Y, Shimokata H. Refractive errors and factors associated with myopia in an adult Japanese population. Jpn J Ophthalmol. 2003 Jan-Feb;47(1):6-12. doi: 10.1016/s0021-5155(02)00620-2. PMID 12586171
- [Background] Vitale S, Sperduto RD, Ferris FL 3rd. Increased prevalence of myopia in the United States between 1971-1972 and 1999-2004. Arch Ophthalmol. 2009 Dec;127(12):1632-9. doi: 10.1001/archophthalmol.2009.303. PMID 20008719
- [Background] Resnikoff S, Pascolini D, Mariotti SP, Pokharel GP. Global magnitude of visual impairment caused by uncorrected refractive errors in 2004. Bull World Health Organ. 2008 Jan;86(1):63-70. doi: 10.2471/blt.07.041210. PMID 18235892
- [Background] Wu PC, Tsai CL, Wu HL, Yang YH, Kuo HK. Outdoor activity during class recess reduces myopia onset and progression in school children. Ophthalmology. 2013 May;120(5):1080-5. doi: 10.1016/j.ophtha.2012.11.009. Epub 2013 Feb 22. PMID 23462271
- [Background] Si JK, Tang K, Bi HS, Guo DD, Guo JG, Wang XR. Orthokeratology for myopia control: a meta-analysis. Optom Vis Sci. 2015 Mar;92(3):252-7. doi: 10.1097/OPX.0000000000000505. PMID 25599338
- [Background] Cooper J, O'Connor B, Watanabe R, Fuerst R, Berger S, Eisenberg N, Dillehay SM. Case Series Analysis of Myopic Progression Control With a Unique Extended Depth of Focus Multifocal Contact Lens. Eye Contact Lens. 2018 Sep;44(5):e16-e24. doi: 10.1097/ICL.0000000000000440. PMID 29053555